CLINICAL TRIAL: NCT02531165
Title: Comparison of Analgesia With Fentanyl and Morphine on Platelet Inhibition After Pre-hospital Ticagrelor Administration in Patients With ST-segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Platelet Inhibition After Pre-hospital Ticagrelor Using Fentanyl Compared to Morphine in Patients With ST-segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Acronym: PERSEUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Dr Juan F. Iglesias, MD, MD, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR14-10591
Record Dates: First submitted 2015-08-18; First posted 2015-08-24 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2018-02

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Fentanyl; Morphine; Ticagrelor; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Morphine (Experimental): * Pre-hospital Ticagrelor 180 mg loading dose orally.
  * Morphine, initial dose: 4-8 mg, additional doses of 2 mg every 5-15 minutes to achieve adequate sedation, if required.
  * Aspirin 500 mg loading dose orally (or intravenously).
  * Unfractioned heparin 5'000 IU loading dose intravenously, additional doses to achieve an ACT >250 sec during PCI are allowed.
  * Primary PCI.
  Interventions: Drug: Morphine; Drug: Ticagrelor; Drug: Aspirin; Drug: Unfractioned Heparin; Procedure: Primary PCI
- Fentanyl (Experimental): * Pre-hospital Ticagrelor 180 mg loading dose orally.
  * Fentanyl, initial dose: 50-100 mcg, additional doses of 25 mcg every 2-5 minutes to achieve adequate sedation, if required.
  * Aspirin 500 mg loading dose orally (or intravenously).
  * Unfractioned heparin 5'000 IU loading dose intravenously, additional doses to achieve an ACT >250 sec during PCI are allowed.
  * Primary PCI.
  Interventions: Drug: Fentanyl; Drug: Ticagrelor; Drug: Aspirin; Drug: Unfractioned Heparin; Procedure: Primary PCI

INTERVENTIONS:
Drug: Fentanyl — Analgesia protocol using Fentanyl (initial dose: 50-100 mcg, additional doses of 25 mcg every 2-5 minutes to achieve adequate sedation, if required).
  Arms: Fentanyl
Drug: Morphine — Analgesia protocol using Morphine (initial dose: 4-8 mg, additional doses of 2 mg every 5-15 minutes to achieve adequate sedation, if required).
  Arms: Morphine
Drug: Ticagrelor — Pre-hospital Ticagrelor loading dose of 180 mg administered orally, followed by 90 mg bid
  Other Names: Brilique
Drug: Aspirin — 500 mg loading dose orally (or intravenously), followed by 100 mg od
Drug: Unfractioned Heparin — 5'000 IU loading dose intravenously, additional doses to achieve an ACT >250 sec during PCI are allowed.
Procedure: Primary PCI — Primary PCI with stent implantation according to the guidelines of the European Society of Cardiology.

SUMMARY:
Prospective, randomized, open-label, single-center, investigator-initiated trial, including patients with ST-segment elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PPCI) within 12 hours of the symptom's onset. The study aims to compare platelet inhibition (pharmacodynamics and pharmacokinetics) of pre-hospital Ticagrelor in patients with STEMI according to two different analgesia protocols using Fentanyl or Morphine.

DETAILED DESCRIPTION:
Consecutive patients with acute STEMI within 12 hours of the symptoms' onset and candidates for PPCI will be screened for inclusion in the study. Eligible patients who require analgesia for the relief of acute chest pain, defined as Visual Analogue Scale ≥3, will be randomized in a 1:1 ratio into one of the two treatment arms to receive analgesia with either Morphine or Fentanyl following administration of a pre-hospital loading dose of Ticagrelor. Randomized patients will undergo primary PCI and managed according to the current guidelines of the European Society of Cardiology. Blood samples (10 ml) will be collected at 0, 1, 2, 4, 6, 12 and 24 hours after the loading dose of Ticagrelor to assess platelet inhibition using the VerifyNow P2Y12 function and the Vasodilator-Stimulated-phosphoprotein Phosphorylation (VASP) assays, plasma concentration of Ticagrelor and its active metabolite (AR-C124910XX) using a validated liquid chromatography/mass spectrometry detection method and the procoagulant action of platelets.

ELIGIBILITY:
Inclusion Criteria:

* Age >18-year-old
* STEMI within 12 hours of symptoms' onset eligible for primary PCI with stent implantation.
* Patient able to give written informed consent.

Exclusion Criteria:

* Contraindication, intolerance or hypersensitivity to Ticagrelor, or any excipients
* Contraindication, intolerance or hypersensitivity to Morphine, Fentanyl, or any excipients
* Active bleeding or bleeding diathesis
* History of intracranial haemorrhage
* Chronic oral anticoagulation treatment
* Previous antiplatelet treatment
* Contraindications to antiplatelet therapy
* Severe renal insufficiency (creatinine clearance <30 mL/min)
* Severe hepatic dysfunction
* Severe chronic obstructive pulmonary disease
* Periprocedural glycoprotein IIb/IIIa inhibitors administration
* Relevant haematological disease
* Patient who is currently, plans, or has been enrolled in another clinical study involving use of an investigational drug or device within the prior 30 days.
* If female, patient pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-09; Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
Residual platelet reactivity (PR) by Platelet Reactivity Units (PRU) | 2 hours after loading dose of Ticagrelor

SECONDARY OUTCOMES:
Residual PR by PRU | 0, 1, 4, 6, 12 and 24 hours after the loading dose of Ticagrelor
High on Treatment Platelet Reactivity (HTPR) rates | 0, 1, 2, 4, 6, 12 and 24 hours after the loading dose of Ticagrelor
Peak plasma concentration (Cmax) of Ticagrelor and AR-C124910XX | at 1, 2, 4, 6 and 12 hours
Time to peak plasma concentration (tmax) of Ticagrelor and AR-C124910XX | at 1, 2, 4, 6 and 12 hours
Area under the plasma concentration-time curve of Ticagrelor | at 1, 2, 4, 6 and 12 hours
Proportion of patients with 70% or greater resolution of the ST-segment elevation before PCI | at 2 hours
Proportion of patients without Thrombolysis in Myocardial Infarction flow grade 3 in the infarct-related artery at initial angiography | at 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Juan F. Iglesias, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Iglesias JF, Valgimigli M, Carbone F, Lauriers N, Giorgio Masci P, Degrauwe S. Effects of Fentanyl Versus Morphine on Ticagrelor-Induced Platelet Inhibition in Patients With ST-Segment Elevation Myocardial Infarction: The PERSEUS Randomized Trial. Circulation. 2020 Dec 22;142(25):2479-2481. doi: 10.1161/CIRCULATIONAHA.120.049287. Epub 2020 Dec 21. No abstract available. PMID 33347326
- [Derived] Degrauwe S, Roffi M, Lauriers N, Muller O, Masci PG, Valgimigli M, Iglesias JF. Influence of intravenous fentanyl compared with morphine on ticagrelor absorption and platelet inhibition in patients with ST-segment elevation myocardial infarction undergoing primary percutaneous coronary intervention: rationale and design of the PERSEUS randomized trial. Eur Heart J Cardiovasc Pharmacother. 2019 Jul 1;5(3):158-163. doi: 10.1093/ehjcvp/pvy031. PMID 30101278